Resilience Program Pilot PI: IT Croghan, PhD Mayo Clinic – NCT04536376

## First Responder Resiliency Program for Health Care Professionals During a Pandemic

Analysis

NCT04536376

12/15/2020

Resilience Program Pilot PI: IT Croghan, PhD Mayo Clinic – NCT04536376

## **General Study Information**

Principal Investigator: Ivana T. Croghan, PhD and Brent A. Bauer, MD

Study Title: First Responder Resiliency Program for Health Care Professionals During a Pandemic

Protocol version number and date: Version 4, December 15, 2020

## **Data Analysis**

**Power Statement:** The sample size for this pilot investigation (N=10) was established after considering both the statistical implications and the amount of project effort and resources required to recruit and study this unique patient population.

**Data Analysis Plan:** Data related to subject recruitment will be summarized, including the frequency of calls and the reasons for failing screening criteria. In all cases, data will be summarized using mean  $\pm$  SD for continuous variables and frequency percentages for nominal variables. Treatment adherence will be quantified for each individual by calculating the percentage of sessions attended. The percentage of subjects who discontinue study participation and the reasons for discontinuing study participation will be summarized.

Patient demographics will be summarized using descriptive statistics. Changes in resilience, stress and sleep will be calculated using a paired t test. In all cases, two-tailed p-values  $\leq 0.05$  will be considered statistically significant.